CLINICAL TRIAL: NCT02399787
Title: Geneexpression as a Marker of Embryo Viability
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Kirstine Kirkegaard, post doc, University of Aarhus
Other Study IDs: 1-10-72-382-13
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- infertile patients: Infertile patients with more than 5 oocytes retrieved and no endometriosis
  Interventions: Other: blastocyst biopsy

INTERVENTIONS:
Other: blastocyst biopsy — Performed on day 5

SUMMARY:
The aim of the post doc project is investigate which genes regulate implantation in order to analyze specific proteins and microRNA in the spent culture media with the long-term goal of developing a non-invasive method of embryo assessment and selection. This will be achieved by conducting a targeted NGS analysis, based on list obtained from a non-published pilot study. When further validated by q-PCR, the expression of specific microRNAs known to influence the final list of genes will be analyzed in the spent culture media and the protein products of the genes recovered from the media will be quantified. The level of specific microRNAs and proteins will be related to aneuploidy and implantation potential. If the level of specific microRNA and/or proteins correlates with pregnancy, the study will form the basis for developing a clinical applicable precise method of improved embryo selection and thus improved IVF treatment.

ELIGIBILITY:
Inclusion Criteria:

* >5 oocytes retrieved

Exclusion Criteria:

* endometriosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infertile women
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
gene expression | 2 years
  the expression of specific microRNAs known to influence the final list of genes will be analyzed in the spent culture media and the protein products of the genes recovered from the media will be quantified. The level of specific microRNAs and proteins will be related to aneuploidy and implantation potential. If the level of specific microRNA and/or proteins correlates with pregnancy, the study will form the basis for developing a clinical applicable precise method of improved embryo selection and thus improved IVF treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Fertility Clinic, Aarhus University Hospital, Skejby, Aarhus, Denmark

REFERENCES:
- See also: publication of results — https://pubmed.ncbi.nlm.nih.gov/32681282/